CLINICAL TRIAL: NCT05520567
Title: A Phase 1/2, Multicenter, Open-Label, Randomized Dose Ranging and Expansion Study of the Combination of Gilteritinib, Venetoclax and Azacitidine in Patients With Newly Diagnosed FLT3 Mutated Acute Myeloid Leukemia (AML) Not Eligible for Intensive Induction Chemotherapy
Brief Title: A Study of Gilteritinib, Venetoclax and Azacitidine as a Combined Treatment for People Newly Diagnosed With Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2215-CL-0203
Record Dates: First submitted 2022-08-26; First posted 2022-08-30 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia (AML); FLT3-mutated Acute Myeloid Leukemia
Keywords: Cancer; Acute Myeloid Leukemia; AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasms | interventions — gilteritinib; venetoclax; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Ranging Cohort (Phase 1) (Experimental): Participants will receive daily dose of gilteritinib and venetoclax for 28 days, and azacitidine for 7 days in each 28-day cycle.
  Interventions: Drug: Gilteritinib; Drug: Venetoclax; Drug: Azacitidine
- Dose Expansion Cohort (Phase 2) (Experimental): Participants will receive daily dose of gilteritinib, venetoclax, and azacitidine at an optimized dose established from dose ranging cohort (Phase 1)
  Interventions: Drug: Gilteritinib; Drug: Venetoclax; Drug: Azacitidine

INTERVENTIONS:
Drug: Gilteritinib — Oral
  Other Names: ASP2215; XOSPATA®
Drug: Venetoclax — Oral
  Other Names: ABT199; Venclexta
Drug: Azacitidine — Subcutaneous injection or intravenous infusion

SUMMARY:
People with acute myeloid leukemia (AML) are usually treated with chemotherapy. Some people with AML have a changed FLT3 gene which causes leukemia cells to grow faster. Therefore, chemotherapy is less suitable to treat AML in people with the changed FLT3 gene.

Gilteritinib, given with venetoclax and azacitidine, is a potential new treatment for people with AML with the changed FLT3 gene. They cannot have chemotherapy due to old age or other conditions. Before these combined 3 medicines are available as a treatment, the researchers need to understand how they are processed by and act upon the body when given together. In this study, they do this to find a suitable dose for venetoclax and to check for potential medical problems from the treatment.

In this study, people newly diagnosed with AML who have the changed FLT3 gene and cannot have chemotherapy can take part.

The main aims of this study are: to find suitable doses of gilteritinib, venetoclax and azacitidine as a combined treatment; to learn how they are processed by and act upon the body; to learn the remission rate; to check for medical problems during this treatment.

In the study, people will visit the study clinic many times. The first visit is to check if they can take part. People will be asked about their medical history, have a medical examination, and have their vital signs checked. Also, they will have an ECG to check their heart rhythm and have some blood and urine samples taken for laboratory tests. They will have a chest X-ray and a bone marrow sample will be taken. The changed FLT3 gene will be confirmed, either by the bone marrow or a blood sample.

This study will be in 2 phases.

In Phase 1, different small groups of people will take venetoclax tablets containing lower to higher doses in the combined treatment. The doses of gilteritinib and azacytidine will be unchanged. This is done to find a suitable dose of venetoclax to use in phase 2 of the study. People will take tablets of gilteritinib and venetoclax once a day on a 28-day cycle. They will be given azacytidine as an infusion or an injection just under the skin. This will be for 7 days at the beginning of each 28-day cycle. They will continue cycles of treatment throughout this phase of the study.

In Phase 2, more people newly diagnosed with AML with the changed FLT3 gene will take part. They will be treated with the suitable doses of the combined treatment worked out from Phase 1. Treatment will be on a 28-day cycle. People will continue on cycles of treatment throughout this phase of the study.

Researchers will work out the remission rate from this phase of the study. In each phase of the study, people can continue with up to 12 cycles of treatment if they can manage any medical problems. People will visit the study clinic many times during their first treatment cycle, and less often during the next cycles. During these visits, medical problems will be recorded and some blood samples will be taken for laboratory tests. On some visits, people will also have their vital signs checked. Bone marrow samples will be taken during cycle 1, and at the beginning of cycle 3. More samples will be taken during the study from people who are not in remission.

When people have finished treatment, those who have responded well to treatment and are in remission will be invited to continue with up to 24 more cycles of gilteritinib plus azacitidine.

All people taking part in the study will visit the study clinic for an end-of-treatment visit. During this visit, medical problems will be recorded and some blood samples will be taken for laboratory tests. People will have a medical examination, an ECG, and will have their vital signs checked. Also, a bone marrow sample will be taken. There will be a follow-up visit 30 days later to check for medical problems. Then people will visit the clinic or get a phone call every 3 months for up to 3 years. This is to give an update on their current treatment for AML.

Some people can have a stem cell transplant during the study if they meet certain study rules. They will pause their study treatment during the stem cell transplant process and continue study treatment afterwards.

ELIGIBILITY:
Inclusion Criteria

* Participant has a diagnosis of previously untreated Acute Myeloid Leukemia (AML) according to World Health Organization classification as determined by pathology review at the treating institution.
* Participant is positive for FMS-like tyrosine kinase 3 (FLT3) mutation (internal tandem duplication [ITD] and/or tyrosine kinase domain [TKD] [D835/I836] mutation) in bone marrow or whole blood as determined by the central laboratory. A participant with rapidly proliferative disease and unable to wait for the central laboratory results can be enrolled from a local test result.
* Participant is ineligible for intensive induction chemotherapy by meeting at least 1 of the following criteria:

  * Participant is >= 75 years of age with Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2.
  * Participant is >= 18 to 75 years of age and has any of the following comorbidities: ECOG performance status 2 or 3, cardiac history of congestive heart failure requiring treatment or ejection fraction <= 50% or chronic stable angina, known history of diffusion capacity of lung for carbon monoxide (DLCO) <= 65% or forced expiratory volume in the first second (FEVI) <= 65%, creatinine clearance > 30 mL/min to 45 mL/min, calculated by the Cockcroft Gault formula, moderate hepatic impairment with total bilirubin > 1.5 to < 3.0 x upper limit of normal (ULN), any other comorbidity incompatible with intensive chemotherapy during screening and before enrollment.
* Participant must have a projected life expectancy of at least 12 weeks.
* Participant must have adequate organ and bone marrow function prior to enrollment, as specified per protocol's laboratory parameters.
* Participant is suitable for oral administration of study drug (gilteritinib and venetoclax) and is willing/able to swallow oral tablets/capsules.
* Participant with a known history of human immunodeficiency virus (HIV) on effective antiretroviral therapy must have a viral load undetectable for 6 months prior to Cycle 1 Day 1 (C1D1).
* Female participant is eligible to participate if she is not pregnant and at least one of the following conditions apply:

  * Not a woman of childbearing potential (WOCBP) OR
  * WOCBP agrees to follow the contraceptive guidance starting at screening and continue through the study treatment period, and for at least 180 days after the final study regimen administration.

WOCBP must have a negative pregnancy test during screening.

* Female participant must agree not to breastfeed starting at screening, throughout the study treatment period and for 60 days after the last dose of the study treatment regimen.
* Female participant must not donate ova starting at screening, throughout the study treatment and for 180 days after the last dose of the study treatment regimen.
* Male participant with female partner(s) of childbearing potential must agree to use contraception starting at screening and continue through the study treatment, and for at least 120 days after the last dose of the study treatment regimen.
* Male participant must not donate sperm starting at screening, throughout the study treatment and for 120 days after the last dose of the study treatment regimen. (Venetoclax may cause a decrease in spermatogenesis. Male participant considering preservation of fertility should bank sperm before initiating treatment with venetoclax.)
* Male participant with a pregnant or breastfeeding partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy or time partner is breastfeeding throughout the treatment period, and for 120 days after the final study drug administration.
* Participant agrees not to participate in another interventional study while on treatment in this study.

Exclusion Criteria:

* Participant with the following conditions:

  * Acute promyelocytic leukemia (APL)
  * Active, symptomatic central nervous system (CNS) involvement with AML
  * History of myeloproliferative neoplasm (MPN), including myelofibrosis, essential thrombocythemia, polycythemia vera, chronic myeloid leukemia (CML) with or without BCR-ABL1 translocation or AML with BCR-ABL1 translocation
* Participant previously treated with CAR-T cell therapy for AML or MDS. Exceptions for prior treatment of AML are (i.e., the following treatments are allowed):

  * Hydroxyurea for increased blast count (No washout period required. It can be continued throughout the first cycle of therapy).
  * Leukapheresis for leukocytosis (No washout period required. It can be continued during the study).
  * Preemptive treatment with retinoic acid prior to exclusion of APL < 7 days.
* Participant who is receiving treatment with any other investigational agents.
* Participant requires treatment with concomitant drugs that are strong or moderate inducers of cytochrome P450 (CYP)3A or P glycoprotein (P-gp) during study treatment.
* Participant who has consumed grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges) or starfruit <= 3 days prior to C1D1.
* Participant with a cardiovascular disability status of New York Heart Association (NYHA) Class >= 3.
* Participant with mean QTcF > 450 msec at screening based on local reading performed in triplicate.
* Participant with a history of Long QT Syndrome at screening.
* Participant has been diagnosed with another malignancy within 2 years prior to screening for the study, with the following exceptions:

  * Adequately treated in situ carcinoma of the cervix uteri or carcinoma in situ of breast;
  * Basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin;
  * Previous malignancy confined and surgically resected (or treated with other modalities) with curative intent
  * Participants who are on maintenance therapy for malignancies with no evidence of active malignancy for >= 2 years and the maintenance therapy can be discontinued.
* Participant who has an uncontrolled intercurrent illness including, but not limited to any of the following conditions:

  * Uncontrolled hypertension
  * Active, uncontrolled infection (viral, bacterial or fungal): An infection controlled with an approved or closely monitored antibiotic/antifungal treatment is allowed.
  * Symptomatic, congestive heart failure
  * Unstable angina pectoris
  * Chronic respiratory disease that requires continuous oxygen
  * Psychiatric illness/social situations that would limit compliance with study requirements
  * Any other illness or condition that would interfere with study compliance or would compromise the participant's safety or study endpoints, including any contraindications to gilteritinib, azacitidine or venetoclax listed in the country package insert.
* Participant who has gastrointestinal disorders, malabsorption or other abnormalities that would interfere with absorption of the oral study drug.
* Participant has active hepatitis B or C or other active hepatic disorder.

  * Participant with positive hepatitis B surface antigen (HBsAg) or detectable hepatitis B virus (HBV) deoxyribonucleic acid (DNA) are not eligible.
  * Participant with negative HBsAg, positive hepatitis B core antibody and negative hepatitis B surface antibody will be eligible if HBV DNA is undetectable.
  * For participant with a known history of chronic HBV infection, the HBV viral load must be undetectable on suppressive therapy, if indicated, to be eligible for this study.
  * Participant with antibodies to hepatitis C virus (HCV) will be eligible if hepatitis C ribonucleic acid (RNA) viral load is undetectable.
  * Participant with a known history of HCV infection must have been treated and cured to be eligible for this study. Participants with HCV infection who are currently on treatment are eligible if they have an undetectable HCV viral load.
* Participant has had major surgery within 4 weeks prior to the first study dose.
* Participant has a known or suspected hypersensitivity to gilteritinib, azacitidine or venetoclax or any components of the formulations used.
* Participant with recent positive test for SARS-CoV-2 ( or diagnosed with COVID-19) and no follow up test with negative result cannot be enrolled. Participant with contact to persons with COVID-19 and participants with signs and symptoms for COVID-19 infection must be tested before enrolling.
* Participant who requires concomitant treatment with a strong or moderate P-gp or CYP3A iinhibitor, with the exception of posaconazole, for antifungal prophylaxis during cycle 1 of the Dose Ranging Phase (phase 1). Note: Posaconazole is the only strong CYP3A inhibitor antifungal allowed during the cycle 1 DLT evaluation period. Post-DLT evaluation period, other antifungals including strong or moderate CYP3A inhibitors are allowed throughout the study.
* Participant does not have any of the following mutations:

FLT3-ITD, FLT3-TKD/D835 or FLT3-TKD/I836.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-01-31 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Dose Limiting Toxicities (DLTs) | Up to 42 Days
  A DLT is defined as any of the events meeting DLT criteria that occur with the first dose on Cycle 1 Day 1 (C1D1) and that is considered to be possibly or probably related to the study treatment regimen.
Number of Participants with Adverse Events (AEs) | Up to 49 months
  An AE is any untoward medical occurrence in a patient or clinical study participant temporally associated with the use of study investigational product (IP), whether or not considered related to the study IP.
  An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study IP. This includes events related to the comparator and events related to the (study) procedures.
Number of Participants with Serious AEs (SAEs) | Up to 49 months
  An SAE is defined as any untoward medical occurrence that, at any dose:
  * results in death
  * is life threatening
  * requires inpatient hospitalization or prolongation of existing hospitalization
  * results in persistent or significant disability/incapacity
  * is a congenital anomaly/birth defect
  * other situations where medical or scientific judgment should be exercised in deciding whether SAE reporting is appropriate in other situations such as important medical events that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed above. These events should usually be considered serious.
Number of Participants with laboratory value abnormalities and/or AEs | Up to 48 months
  Number of participants with potentially clinically significant laboratory values.
Number or Participants with electrocardiogram (ECG) abnormalities and/or AEs | Up to 48 months
  Number of participants with potentially clinically significant ECG values.
Number of Participants with vital sign abnormalities and/or AEs | Up to 48 months
  Number of participants with potentially clinically significant vital sign values.
Number of Participants with physical exam abnormalities and/or AEs | Up to 48 months
  Number of participants with potentially clinically significant physical exam values.
Number of Participants at each grade of the Eastern Cooperative Oncology Group (ECOG) performance status scores | Up to 48 months
  The ECOG scale will be used to assess performance status. Grades range from 0 (fully active) to 5 (dead). Negative change scores indicate an improvement. Positive scores indicate a decline in performance.
Percentage of Participants with Complete Remission (CR) | Up to 24 months
  CR rate is defined as the number of participants who achieve the best response of CR divided by the number of participants in the analysis population.
  CR is defined as participants having bone marrow regenerating normal hematopoietic cells and achieve a morphologic leukemia-free state and must have bone marrow blasts < 5% by morphological examination, absolute neutrophil count (ANC) > 1 x 10^9/L, platelet count > 100 x 10^9/L, and an absence of leukemic blasts in the peripheral blood by morphological examination. There should be no evidence of extramedullary disease. Other participants who do not relapse on study are considered nonevents and censored at the last
Pharmacological activity by Plasma Inhibitory Activity Assay (PIA) | Up to 2 months
  Inhibition of FLT3 phosphorylation after drug treatment will be determined relative to pretreatment phosphorylated FLT3 levels in participants to assess the relationship with gilteritinib dose. Phosphorylated FLT3 will be measured by plasma inhibitory activity (PIA) assay.
Pharmacokinetics (PK) of ASP2215 in plasma: concentration | Up to 6 months
  Concentration will be recorded from the PK plasma samples collected.

SECONDARY OUTCOMES:
Percentage of Participants with Complete Remission and Complete Remission with Partial Hematological Recovery (CR/CRh) rate | Up to 24 months
  The CR/CRh rate is defined as the number of participants who achieved either CR or CRh at any of the post baseline visits divided by the number of participants in the analysis population.
Percentage of Participants with Composite Complete Remission (CRc) | Up to 24 months
  CRc rate is defined as the number of participants who achieve the best response of CRc divided by the number of participants in the analysis population.
Duration of Remission (DOR) | Up to 24 months
  Duration of remission includes duration of CRc, CR, CR/CRh, CRh, complete remission with incomplete hematologic recovery (CRi), complete remission with incomplete platelet recovery (CRp).
  Duration of CRc is defined as the time from the date of first CRc until the date of confirmed relapse or death due to any cause for participants who achieve CRc. Participants without confirmed relapse or death will be censored at their last relapse-free disease assessment date. The duration of CR, CR/CRh, CRh, CRp or CRi is defined similarly as duration of CRc.
Duration of Overall Survival (OS) | Up to 24 months
  OS is defined as the time from the date of enrollment until the date of death from any cause. For a participant who is not known to have died by the end of study follow-up, OS is censored at the date of last contact.
Duration of Event free survival (EFS) | Up to 24 months
  EFS is defined as the number of days from the date of enrollment to the date of earliest evidence of relapse, treatment failure, or death.
Pharmacokinetics (PK) of ASP2215 in plasma: area under the plasma concentration-time curve during a dosage interval (AUCtau) | Up to 6 months
  AUCtau will be recorded from the PK plasma samples collected.
PK of ASP2215 in plasma: maximum observed concentration (Cmax) | Up to 6 months
  Cmax will be recorded from PK plasma samples collected.
PK of ASP2215 in plasma: pre-dose trough concentration (Ctrough) | Up to 6 months
  Ctrough will be recorded from PK plasma samples collected.
PK of ASP2215 in plasma: area under the curve from time 0 to the time of the last measurable concentration (AUClast) | Up to 6 months
  AUClast will be recorded from PK plasma samples collected.
PK of ASP2215 in plasma: time to Cmax (tmax) | Up to 6 months
  tmax will be recorded from PK plasma samples collected.
Number of participants with negative minimal residual disease (MRD) status | Up to 48 months
  MRD testing will be performed on left over bone marrow samples taken at different time points during the study, and at end of treatment.
Transplantation rate | 24 months
  Transplantation rate is defined as the percentage of participants undergoing hematopoietic stem cell transplantation (HSCT) during the study treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (20):
- United States (20):
  - City of Hope Nat'l Medical Center, Duarte, California
  - Univ. of California - Irvine, Irvine, California
  - UCLA Medical Center, Los Angeles, California
  - Sarah Cannon Research Institute, Denver, Colorado
  - Memorial Cancer Institute, Pembroke Pines, Florida
  - University of Chicago, Chicago, Illinois
  - Robert H. Lurie Comprehensive Cancer Center, Chicago, Illinois
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Roswell Park Cancer Institute, Buffalo, New York
  - Weill Cornell Medical College, New York, New York
  - Motefiore-Einstein Center for Cancer Care, The Bronx, New York
  - Novant Health, Winston-Salem, North Carolina
  - Ohio State University, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania-Abramson CCC-Dept. of Hem Onc, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - The University of Texas MD, Houston, Texas
  - The Medical College of Wisconsin- Froedtert Hospital, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/